CLINICAL TRIAL: NCT03380065
Title: Comparison of Two Protocols for Deflation of Radial Band Following Coronary Procedures Via the Radial Route
Brief Title: Comparison of Two Protocols for Deflation of Radial Band Following Coronary Procedures Via the Radial Artery
Acronym: SQUARE1
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan Qaboos University (Other)
Responsible Party: Principal Investigator, SUNIL NADAR, Senior Consultant, Sultan Qaboos University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SQUARE1
Record Dates: First submitted 2017-12-11; First posted 2017-12-20 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Coronary Artery Disease; Radial Artery Injury
Keywords: coronary angiogram; radial artery
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Late deflation of TR band (Active Comparator): 1. first 3ml of air removed from the TR band after TWO hour of sheath removal. Then, 3ml of air removed every 15minutes.
  2. Observe for any bleeding or hematoma. During every deflation, if any bleeding or hematoma is noticed then 3ml of air is pushed back into the device until bleeding stops. Then wait for another 15minutes for the next deflation.
  Interventions: Device: Late deflation of TR band
- Early deflation of TR band (Active Comparator): 1. First 2ml of air is removed from the TR band ONE hour after sheath removal. Then, 2ml of air is removed every 30minutes.
  2. Observe for any bleeding or hematoma. During every deflation, if any bleeding or hematoma is noticed then push the 2ml of air back into the device until bleeding stops. Then wait for another 30minutes for the next deflation.
  Interventions: Device: Early deflation of TR band

INTERVENTIONS:
Device: Late deflation of TR band — 1. First 3ml of air is removed after TWO hour of sheath removal. Then, 3ml of air is removed every 15minutes.
  2. Observe for any bleeding or hematoma. During every deflation, if any bleeding or hematoma is noticed then 3ml of air is pushed back into the device until bleeding stops. Then a gap of 15minutes is observed for the next deflation.
  Other Names: Late deflation
  Arms: Late deflation of TR band
Device: Early deflation of TR band — 1. First 2ml of air is removed from the band ONE hour after sheath removal. Then, 2ml of air is removed every 30minutes.
  2. Observe for any bleeding or hematoma. During every deflation, if any bleeding or hematoma is noticed then 2ml of air should be pushed back into the device until bleeding stops. Then wait for another 30minutes for the next deflation.
  Arms: Early deflation of TR band

SUMMARY:
Coronary angiography is now mainly performed via the radial route rather than the femoral route. At the end of the procedure, the sheath is removed and a band is inflated to obtain hemostasis. The air in the band is then deflated at regular intervals. Currently there are different protocols for deflation of the band, but none of these have been studied with regards to patient comfort and time of deflation, and potential complications such as bleeding. Here in this study the investigators wish to compare two such protocols of band deflation and assess the levels of patient comfort and time to discharge with two widely used protocols.

DETAILED DESCRIPTION:
Coronary angiography is a procedure by which the anatomy of the coronary arteries are studied. It can be done either via the radial artery approach or the femoral artery approach. Currently most centers use the radial artery approach due to the lower risk of access site bleeding as compared to the femoral artery approach. In addition, the radial approach allows earlier patient mobilisation after the procedure.

Once the sheath, through which the procedure is done, is removed, a special air filled band is used to compress the artery to prevent bleeding. This involves filling the band with around 18 ml of air and then releasing the air at periodic intervals. There are however no set protocols for the removal of air and literature often suggests varying protocols. However what the protocols try to achieve is proper hemostasis, with low incidence of radial artery occlusion. In addition to these, patient comfort and safety along with staff ease of use is important. Some protocols involve frequent deflations which might be more tedious for the nurses, but more comfortable for patients whilst others might be easier for the staff (due to longer intervals), but more uncomfortable for the patients. However, there are no studies that actually compare these protocols

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing coronary procedures via the radial route

Exclusion Criteria:

* Those below the age of 18 and those unable to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2018-01-30 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-20 (Actual)

PRIMARY OUTCOMES:
Total deflation time | 2 hours
  To see how quickly the band can be removed in each arm

SECONDARY OUTCOMES:
Staff satisfaction | 2 hours
  using a visual analogue scale (from 1-10 where 1 is totally dissatisfied and 10 is completely satisfied
Patient satisfaction | 2 hours
  using a visual analogue scale (from 1-10 where 1 is extremely painful and uncomfortable and 10 is totally unpainful and comfortable

CONTACTS AND LOCATIONS:
Overall Officials: Adil Riyami, MD, Principal Investigator — Sultan Qaboos University
Locations (1):
- Sultan Qaboos University Hospital, Muscat, Alkhod, Oman

IPD SHARING:
Plan to Share IPD: Undecided
The data regarding the time of band deflations and patient and staff satisfaction scores